CLINICAL TRIAL: NCT05677438
Title: A Phase 2, Randomized, Double-blind, Multi-center, Parallel-group Trial to Evaluate the Efficacy and Safety of CKD-498 in Female Patients With Androgenetic Alopecia
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of CKD-498 in Female Patients With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A128_01AGA2211
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenetic Alopecia; CKD-498
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test Group1 (Experimental)
  Interventions: Drug: CKD-498 dose#1; Drug: Placebo of CKD-498 dose#2; Drug: Placebo of CKD-498 dose#3
- Test Group2 (Experimental)
  Interventions: Drug: CKD-498 dose#2; Drug: Placebo of CKD-498 dose#1; Drug: Placebo of CKD-498 dose#3
- Test Group3 (Experimental)
  Interventions: Drug: CKD-498 dose#3; Drug: Placebo of CKD-498 dose#1; Drug: Placebo of CKD-498 dose#2
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo of CKD-498 dose#1; Drug: Placebo of CKD-498 dose#2; Drug: Placebo of CKD-498 dose#3

INTERVENTIONS:
Drug: CKD-498 dose#1 — oral, once daily, 24 weeks
  Arms: Test Group1
Drug: CKD-498 dose#2 — oral, once daily, 24 weeks
  Arms: Test Group2
Drug: CKD-498 dose#3 — oral, once daily, 24 weeks
  Arms: Test Group3
Drug: Placebo of CKD-498 dose#1 — oral, once daily, 24 weeks
  Arms: Placebo Group; Test Group2; Test Group3
Drug: Placebo of CKD-498 dose#2 — oral, once daily, 24 weeks
  Arms: Placebo Group; Test Group1; Test Group3
Drug: Placebo of CKD-498 dose#3 — oral, once daily, 24 weeks
  Arms: Placebo Group; Test Group1; Test Group2

SUMMARY:
This is a multi-centers, randomized, double-blind, parallel-group, Phase 2 Trial to evaluate the efficacy and safety of CKD-498 in female patients with Androgenetic Alopecia

DETAILED DESCRIPTION:
Participants were randomly assigned in a 1:1:1:1 ratio to the following group: 3 dose of CKD-498 and Placebo. The patients are prescribed oral administration of the appropriate IP daily (3 tablets: actual medication and placebo) for 24 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Female of age 19-54 years
* Clinical Diagnosis of Androgenetic Alopecia
* Written informed consent

Key Exclusion Criteria:

* Other types of Alopecia or other diseases that can cause hair loss
* Clinically significant scalp disease such as seborrheic dermatitis or psoriasis
* Clinically significant hepatic disease, thyroid disease, or mental illness, as determined by the Investigator
* Women who are pregnant or breastfeeding
* Women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the last dose of study drug

Ages: 19 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Total number of hair Changes | Baseline, Week 24
  from Baseline at Week24 of total number of hair changes

CONTACTS AND LOCATIONS:
Overall Officials: ChangHun Huh, MD, PhD., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No